CLINICAL TRIAL: NCT01523535
Title: Repeated Challenge of Insufficient Sleep: Effects on Endothelial Function
Brief Title: Repeated Challenge of Insufficient Sleep: Endothelial Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Janet M Mullington, PhD, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010P000365; R01HL106782 (NIH)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2018-07

CONDITIONS: Repeated Short Sleep Schedule

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants were randomized to condition. Vascular reactivity testing was performed by operator who was blind to condition and outcomes assessment from that testing was also blind.
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal sleep (Placebo Comparator): Subjects have 8 hours of sleep opportunity per night
  Interventions: Behavioral: repeated cycles of short sleep
- cycles of sleep restriction (Experimental): subjects are exposed to bouts of reduced sleep duration. The sleep loss is the intervention (experimental challenge).
  Interventions: Behavioral: repeated cycles of short sleep

INTERVENTIONS:
Behavioral: repeated cycles of short sleep — - 3 nights of 4 hours of sleep followed by a single recovery night of 8 hours; repeated for 4 cycles

SUMMARY:
The 24-hour-a-day, 7-day a week, work-world arrived within our lifetimes, and is here to stay. Americans are working more and more, frequently at multiple jobs. The pattern of short sleep during the week followed by attempts to recover on the weekend is in common practice, but we know little of the associated health risks. What is the cost in terms of increasing known risk markers for cardiovascular disease, of repeated nights of insufficient sleep, and is this cost compounded with repetition, without adequate recovery? Evidence is accumulating to suggest that short sleep duration is linked to the development of metabolic and inflammation-associated diseases, such as cardiovascular disease. Mechanisms involved in the development of cardiovascular disease include impaired vascular function and inflammation. The current proposal is designed to investigate the effects of repeated periods of short nocturnal sleep duration in 4 cycles (each cycle consisting of 3 nights of 4 hours of sleep opportunity per night), and each cycle of short sleep followed by a single night of recovery sleep. Vascular reactivity will be assessed using brachial artery flow mediated dilation, and microcirculatory vasodilation will be assessed using perfusion imaging techniques. The dependence of IL-6 and sVCAM-1 as measured in peripheral circulation, on vascular function, will also be investigated.

DETAILED DESCRIPTION:
Due to work, family, social and community obligations, millions of Americans cut back on sleep for several nights in a row before having an opportunity to catch up. When the opportunity does arise, it may only be for a single night, before the cycle of insufficient sleep repeats. This study investigated what happens to human biology when insufficient sleep becomes chronic and opportunities for recovery sleep are intermittent. It also investigated recovery sleep itself, and the biological processes involved in reversing the effects of an accumulated sleep deficit due to insufficient sleep duration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Regular sleep-wake schedule

Exclusion Criteria:

* Diseases or medical conditions, including sleep disorders
* Current smoking
* Pregnant or nursing
* Recent time zone travel or shift work
* Regular medication use
* High blood pressure

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Vascular reactivity | 22 days

SECONDARY OUTCOMES:
Inflammation | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Mullington, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No